CLINICAL TRIAL: NCT04898634
Title: A Phase 1 Study of JNJ-78278343, a T-Cell-Redirecting Agent Targeting Human Kallikrein 2 (KLK2), for Advanced Prostate Cancer
Brief Title: A Study of JNJ-78278343, a T-Cell-Redirecting Agent Targeting Human Kallikrein 2 (KLK2), for Advanced Prostate Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CR108958; 78278343PCR1001 (Other: Janssen Research & Development, LLC); 2020-005970-83 (EudraCT Number); 2023-506585-31-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2021-05-20; First posted 2021-05-24 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostatic Neoplasms
Keywords: Metastatic castration-resistant prostate cancer (mCRPC); Advanced prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- JNJ-78278343 (Experimental): Participants will receive JNJ-78278343. The dose levels will be escalated based on the dose limiting toxicities (DLT) evaluation by the study evaluation team (SET) in Part 1 (dose escalation). In Part 2 (dose expansion), participants will receive JNJ-78278343 at recommended phase 2 dose (RP2D) as determined in Part 1. Participants who are still on study treatment (i.e., who are in Treatment Phase) at the time of the long term extension (LTE) will continue to receive study treatment until they reach a reason for discontinuation of treatment or until further notification by the sponsor of a different means for continued supply of study treatment, whichever occurs first.
  Interventions: Drug: JNJ-78278343

INTERVENTIONS:
Drug: JNJ-78278343 — JNJ-78278343 will be administered.

SUMMARY:
The purpose of this study is to determine the recommended phase 2 dose(s) (RP2Ds) of JNJ-78278343 in Part 1 (Dose Escalation) and the safety at the RP2Ds in Part 2 (Dose Expansion).

ELIGIBILITY:
Inclusion Criteria:

* Confirmed adenocarcinoma of the prostate which has spread to other body parts
* Part 1: Prior treatment with at least 1 prior novel androgen receptor (AR)-targeted therapy or chemotherapy
* Measurable or evaluable disease
* Concurrent use of any other anticancer treatment must be discontinued for at least 2 weeks before the first dose of study drug
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Prior surgical removal of testicles; or, for participants who have not undergone surgical removal of testicles, must be receiving ongoing androgen deprivation therapy (ADT) with a gonadotropin releasing hormone analog

Exclusion Criteria:

Disease conditions

* Active central nervous system (CNS) involvement
* Toxicity related to prior anticancer therapy has not adequately recovered

Prior/Concomitant Therapy

* Prior treatment with human kallikrein (KLK) 2-targeted therapy
* Received, or are receiving, medications that suppress the immune system within 3 days prior to the first dose of study drug
* Received or plans to receive any live, attenuated vaccine within 4 weeks prior to the first dose of study drug

Prior/Concurrent Medical Conditions

* Diagnosis of cancer other than prostate cancer within 2 years prior to the first dose of study drug
* Solid organ or bone marrow transplantation
* Major clotting diseases within one month prior to the first dose of study drug
* Active autoimmune disease within 12 months prior to the first dose of study drug
* Active infection
* Major diseases of heart and blood vessels within 6 months prior to the first dose of study drug
* Clinically significant lung diseases
* Active or chronic hepatitis B or hepatitis C infection
* Known positive test result for human immunodeficiency virus (unless stable on antiretroviral therapy with undetectable viral load)
* Any serious underlying medical conditions or other issue that would impair the ability of the participant to receive or tolerate the planned treatment

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 216 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2027-02-10 (Estimated)

PRIMARY OUTCOMES:
Part 1 and 2: Number of Participants With Adverse Events (AEs) | Up to 1 year and 10 months
  An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study.
Part 1 and 2: Number of Participants With AEs by Severity | Up to 1 year and 10 months
  Severity will be graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0. Severity scale ranges from Grade 1 (Mild) to Grade 5 (Death). Grade 1= Mild, Grade 2= Moderate, Grade 3= Severe, Grade 4= Life-threatening and Grade 5= Death related to adverse event. Cytokine release syndrome (CRS) and immune effector cell associated neurotoxicity syndrome (ICANS) will be graded according to the American Society for Transplantation and Cellular Therapy (ASTCT) guidelines.
Part 1: Number of Participants With Dose-Limiting Toxicity (DLT) | Up to 1 year and 10 months
  Number of participants with DLT will be reported. The DLTs are specific adverse events and are defined as any of the following: high grade non-hematologic toxicity, or hematologic toxicity.

SECONDARY OUTCOMES:
Serum Concentration of JNJ-78278343 | Up to 1 year and 10 months
  Serum concentrations of JNJ-78278343 will be determined.
Systemic Cytokine Concentrations | Up to 1 year and 10 months
  Cytokine concentrations will be determined for biomarker assessment.
Serum Prostate Specific Antigen (PSA) Concentration | Up to 1 year and 10 months
  Serum PSA concentration will be measured.
Number of Participants With Anti-JNJ-78278343 Antibodies | Up to 1 year and 10 months
  Serum samples will be analyzed for the detection of anti-JNJ-78278343 antibodies using a validated assay method.
Objective Response Rate (ORR) | Up to 1 year and 10 months
  ORR is defined as the percentage of participants who have a partial response (PR) or better according to the response evaluation criteria in solid tumors (RECIST) version 1.1 response criteria without evidence of bone progression according to prostate cancer working group 3 (PCWG3).
Radiographic Progression-free Survival (rPFS) | Up to 1 year and 10 months
  rPFS is defined as time from the date of first dose of JNJ-78278343 until the date of objective disease progression or death, whichever comes first.
PSA Response Rate | Up to 1 year and 10 months
  PSA response rate is defined as the percentage of participants with a decline of PSA of 50 percent (%) or more from baseline. The maximum reduction from baseline in PSA will also be calculated during the treatment.
Duration of Response (DOR) | Up to 1 year and 10 months
  DOR will be calculated among responders (PR or better) from the date of initial documentation of a response (PR or better) to the date of first documented evidence of progressive disease, as defined in the PCWG3 or RECIST version 1.1 response criteria, or death due to any cause, whichever occurs first.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (17):
- United States (3):
  - Columbia University Medical Center Herbert Irving Pavilion, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Washington, Seattle, Washington
- China (4):
  - Peking University Third Hospital, Beijing
  - Chongqing University Cancer Hospital, Chongqing
  - Sun Yat Sen University Cancer Center, Guangzhou
  - First Affiliated Hospital Of Wenzhou Medical College, Wenzhou
- France (3):
  - Centre Leon Berard, Lyon
  - APHM Hopital Timone, Marseille
  - Institut Gustave Roussy, Villejuif
- Japan (2):
  - National Cancer Center Hospital East, Kashiwa
  - Yokohama City University Medical Center, Yokohama
- Netherlands (2):
  - Antoni van Leeuwenhoek, Amsterdam
  - Erasmus MC, Rotterdam
- Spain (3):
  - Hosp Univ Fund Jimenez Diaz, Madrid
  - Hosp Univ Hm Sanchinarro, Madrid
  - Hosp Virgen de La Victoria, Málaga

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at www.innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency

REFERENCES:
- [Derived] Stein MN, Vinceneux A, Robbrecht D, Doger B, Autio KA, Schweizer MT, Calvo E, Medina L, Van Dongen M, Deville JL, Bernard-Tessier A, Ghosh D, Shotts K, Shen F, Jaiprasart P, Chaudhary R, Wu S, Cartee L, Schnepp R, Gaut D, Lauring J, Wang SC, Villalobos VM, Baldini C. Pasritamig, a First-in-Class, Bispecific T-Cell Engager Targeting Human Kallikrein 2, in Metastatic Castration-Resistant Prostate Cancer: A Phase I Study. J Clin Oncol. 2025 Aug;43(22):2515-2526. doi: 10.1200/JCO-25-00678. Epub 2025 Jun 1. PMID 40450573